CLINICAL TRIAL: NCT01160705
Title: Biomarkers of Response to Taxotere in Hormone-Refractory Prostate Cancer
Brief Title: Biomarkers of Response to Taxotere in HRPC. ICORG 08-08, V2
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 08-08; ICORG-08-08; EU-21044
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; bone metastases; liver metastases; lung metastases; hormone-resistant prostate cancer
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Docetaxel; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: docetaxel
Genetic: RNA analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: circulating tumor cell analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying blood samples in predicting how patients with prostate cancer will respond to treatment with docetaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if mRNA present in circulating tumor cells will help predict response in patients with hormone-refractory prostate cancer treated with docetaxel.
* In parallel with this, based on discoveries made since our protocol was initially submitted to ICORG, here we also propose to analyse serum specimens from these consenting patients for the presence of EC miRNA, mRNA and protein predictive of response to Taxotere.

Secondary

* To develop a predictive model based on the most accurate and sensitive combination of these biomarkers.

OUTLINE: This is a multicenter study.

Treatment Plan:

All patients will be treated with Docetaxel on a weekly, biweekly or three weekly schedule, dose and schedule at the discretion of the treating physician.

Blood samples are collected for biomarker laboratory studies at baseline, every 3-4 weeks during study, and at disease progression or every 12 weeks after completion of study. Samples are analyzed for mRNA via RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following criteria:

1. Patients must, in the opinion of the Investigator, be suitable for treatment with Docetaxel on a weekly, biweekly or three weekly schedule.
2. Patients must be aged 18 years or over.
3. Patients must have histologically or cytologically proven adenocarcinoma of the prostate gland.
4. Patients must have evidence of locally advanced or metastatic disease (e.g. bone, pelvic mass, lymph node, liver or lung metastases).
5. Patients must have had prior treatment with bilateral orchiectomy or other primary hormonal therapy (LHRH-agonist etc.) with evidence of treatment failure.
6. Patients must not have received prior treatment with chemotherapy.
7. Patients must be able to give written informed consent.
8. Prior radiotherapy is allowed.
9. Concomitant use of bisphosphonates is allowed.

Exclusion Criteria:

1. Patients who have received previous cytotoxic therapy for prostate cancer are ineligible.
2. Patients who in the judgement of their treating physician will not be able to receive therapy and follow-up according to the protocol guidelines will be ineligible.
3. Presence of a medical or psychiatric condition, which, in the opinion of the investigator, would potentially pose a risk to the patient by participating in this trial.
4. History of other primary cancer, unless:

   * Curatively resected non-melanomatous skin cancer
   * Other primary solid tumour curatively treated with no known active disease present and no curative treatment for the last year.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hormone refractory Prostate Cancer patients who are due to receive their first treatment with Docetaxel.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2009-11; Primary Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Presence of mRNA in circulating tumor cells as a predictor of response | ongoing

SECONDARY OUTCOMES:
Development of a predictive model | End of trial

CONTACTS AND LOCATIONS:
Overall Officials: Ray McDermott, MD, Principal Investigator — Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital
Locations (5):
- Ireland (5):
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Private Hospital, Dublin